CLINICAL TRIAL: NCT01768377
Title: Comparison of in Intubation With Nerve Block and Intubation With Sedation in Awake Patients in Terms of Efficacy, Complications and Physician's Satisfaction
Brief Title: Comparison of Intubation With Nerve Block and With Sedation in Awake Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130-1928
Record Dates: First submitted 2013-01-01; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Intubation Complication
Keywords: Awake intubation; Nerve block; Sedation; Physician satisfaction
MeSH Terms: interventions — Nerve Block; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation with sedation (Active Comparator): Sedation with midazolam and analgesia with fentanyl
  Interventions: Drug: Fentanyl; Drug: Midazolam
- Intubation with Nerve block (Experimental): Laryngeal plus supraglottic plus intratracheal nerve block plus sedation with midazolam
  Interventions: Drug: Nerve block with Lidocain; Drug: Midazolam

INTERVENTIONS:
Drug: Nerve block with Lidocain — Lidocain 2% topical injection, 0.5 - 1 cc Lidocain 4% topical injection, 3 cc Lidocain 10% topical spray , total dose 50 mg
  Arms: Intubation with Nerve block
Drug: Fentanyl — Fentanyl 2 microgram/Kg BW IV
  Arms: Intubation with sedation
Drug: Midazolam — Midazolam 0.05 mg/kg BW IV infusion

SUMMARY:
The purpose of this study is to compare intubation with nerve block with intubation with sedation in awake patients in terms of efficacy, ease, and the rate of complications and physician satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Candidate for intubation with methods other than RSI
* Age>= 18 years
* Patient or patient's guardian's consent

Exclusion Criteria:

* Need for RSI or crash intubation
* Allergy to Lidocain in block group
* Allergy to opioid drugs in sedation group
* Allergy to midazolam in either group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Time required for intubation in seconds | From start of the intubation attempt for an average of one minutes
  The interval is measured from the time that the healthcare provider attempts intubation until a successful intubation is achieved.

SECONDARY OUTCOMES:
physicians' perception of the difficulty of the procedure | Within an average of 30 minutes after completion of the procedure
  Physicians' perception about the difficulty of the procedure is assessed using a 5-point Likert type scale (ranging from very easy to very difficult)verbally administered to the healthcare provider immediately (within 30 minutes) after completion of the intubation
Number of Participants with Adverse Events | From the start of the procedure until 30 minutes after the procedure is completed
  Number of patients developing any of the following complications (cough, esophageal intubation) from the start of the procedure until 30 minutes after completion of the procedure. This will represent the rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jalili, MD, Study Director — TUMS; Amir Nejati, MD, Principal Investigator — TUMS
Locations (1):
- Imam Khomeini Hospital, Tehran, Tehran Province, Iran